CLINICAL TRIAL: NCT04305067
Title: PRECISE: PancREatic Cancer and Individualised Supervised Exercise: a Feasibility Study
Brief Title: PRECISE: Pancreatic Cancer and Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: Pancreatic Cancer UK (Other); Belfast Health and Social Care Trust (Other)
Responsible Party: Principal Investigator, Gillian Prue, Senior lecturer in chronic illness, Queen's University, Belfast
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: B19/35
Record Dates: First submitted 2020-02-28; First posted 2020-03-12 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Pancreas Adenocarcinoma
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supervised aerobic and resistance exercise (Experimental): 16 weeks of supervised, moderate intensity, aerobic and resistance exercise. Aerobic exercise will be completed supervised, 2 days per week, commencing with a single 10 minute bout and progressing to 30 minutes of continuous aerobic exercise. Resistance exercises will involve whole body activities and commence with 1 set of each exercise (6-12 repetitions) and progress to 3 sets. The resistance exercises will gradually progress in difficulty throughout the program and will utilise daily undulating periodisation
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Exercise programs will be individually tailored to the capabilities of each participant and gradually progressed accordingly. Each patient will be asked to complete one home-based aerobic exercise sessions each week. At baseline, 16 weeks and 3 month followup patients will complete a physical fitness assessment (30 second sit to stand and six minute walking tests) and a range of quality of life questionnaires. Upon completion of the 16 week exercise intervention, patients will be invited to partake in semi-structured interviews to determine the effectiveness of the program and their experience throughout.

SUMMARY:
The purpose of this study is to establish the feasibility of delivering a prescribed, individualised supervised aerobic and resistance exercise programme during adjuvant therapy, to improve survival and reduce symptom burden in pancreatic cancer

DETAILED DESCRIPTION:
Pancreatic ductal adenocarcinoma (PDAC) is the most common malignancy of the pancreas, representing 90% of all pancreatic neoplasms. The late presentation of symptoms and a lack of effective screening methods, means a large proportion (80-90%) are diagnosed with unresectable advanced disease, contributing to an unfavorable prognosis and dismal 5-year survival rate of ~5%. Intensive cancer treatments (i.e. surgery and chemotherapy) have debilitating complications including fatigue, pain and impaired physical function. Therefore, the maintenance of physical function and quality of life are seen as primary treatment goals for pancreatic patients, particularly during adjuvant therapy. Exercise training is emerging as an accepted component of patient care and evidence suggests regular exercise may induce an array of physiological and psychosocial benefits. However, there is a lack of evidence on the feasibility of delivering supervised exercise interventions to individuals with resectable PDAC undergoing adjuvant therapy. This study aims to explore the initial feasibility of delivering a supervised, individualized, and progressive concurrent exercise intervention to individuals with resectable PDAC who are undergoing adjuvant therapy, and provide data required to design a future randomized controlled trials.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* histologically proven pancreatic ductal adenocarcinoma
* complete macroscopic resection (R0 or R1 resection)
* patients recovering from surgery in time for chemotherapy to be delivered with adjuvant intent
* prior malignancy active within the previous 3 years other than locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* deemed medically fit by treating team to participate in exercise programme
* able to provide informed consent.

Exclusion Criteria:

* Macroscopically remaining tumour (R2 resection or tumour node metastasis (TNM) stage IV disease)
* Pre-existing cardiac conditions; Congestive heart failure or recent serious cardiovascular event
* Chest pain while undertaking physical activity
* Any related co-morbidities (diabetes; unstable angina; degenerative neuromuscular disease; mental health disorders; substance abuse)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Feasibility - recruitment: number of participants that agree to participate or are excluded | At baseline
  The number of participants that agree to participate or are excluded
Feasibility - attrition: number of participants that withdraw from the study | At conclusion of the 16 week exercise intervention
  The number of participants that withdraw from the study
Feasibility - adherence to the exercise intervention: percentage of participants adhering to the exercise intervention | At conclusion of the 16 week exercise intervention
  Determine the percentage of participants adhering to the exercise intervention
Feasibility - participant experience: semi-structured interviews | At conclusion of the 16 week exercise intervention
  Determined by qualitative evaluation, using semi-structured interviews to assess experiences, accessibility and acceptability of the exercise intervention

SECONDARY OUTCOMES:
Anthropometric assessment | At baseline, 16 weeks, 3 month follow-up
  Height will be measured in cm and body weight in k, which will be combined to report BMI in kg/m (squared).
Hip and waist circumference analysis | At baseline, 16 weeks, 3 month follow-up
  Hip and waist circumference will be measured in cm.
Functional muscle endurance assessment | At baseline, 16 weeks, 3 month follow-up
  The amount of repetitions achieved during a 30 second sit-to-stand test will be recorded.
Physical fitness assessment | At baseline, 16 weeks, 3 month follow-up
  Distance covered in meters during a six minute walk test will be recorded.
Perceived physical activity levels | At baseline, 16 weeks, 3 month follow-up
  Patients will complete an International Physical Activity Questionnaire (IPAQ-SF). This questionnaire will comprise 4 generic items to obtain comparable health-related physical activity. Patients will detail the number of days, hours and minutes that they undertake (1) vigorous exercise (2) moderate exercise (3) walking exercise and (4) sitting. Total physical activity will be generated and monitored for improvement or decline. Higher reported scores indicate higher levels of self-reported physical activity.
Cancer-related fatigue by questionnaire | At baseline, 16 weeks, 3 month follow-up
  Fatigue will be measured by the Functional Assessment of Cancer Therapy - Fatigue (FACIT-Fatigue) questionnaire. Patients will score several fatigue items over the past 7 days on a scale (0 = not at all; 4 = very much), generating a total (0 - 52) with higher scores linked to greater quality of life.
Patient rated pain by questionnaire | At baseline, 16 weeks, 3 month follow-up
  Pain will be measured using the Brief Pain Inventory (BPI). Pain is scored on a scale 0 - 10, with higher scores indicating higher pain levels.
Well-being by questionnaire | At baseline, 16 weeks, 3 month follow-up
  Quality of life will be measured by the Functional Assessment of Cancer Therapy-Hepatobiliary (FACT-Hep) questionnaire. This questionnaire is scored on a scale of 0 - 4, with 0 indicating not at all, and 4 indicating very much. Higher scores indicate poorer quality of life.
Health related quality of life by questionnaire | At baseline, 16 weeks, 3 month follow-up
  Quality of life will be measured by the EuroQOL Five Dimension Questionnaire (EQ5D). Patients will select a level of difficulty (I have no - I have extreme) on that particular days health for mobility, self-care, usual activities, pain / discomfort and anxiety / depression. Patients will then rate 'how good' or 'how bad' their health is on that day using a 100 point scale (0 = worst health you can imagine; 100 = best health you can imagine).
Health economics | At 16 weeks
  Health resource use will be evaluated by a Health Economics Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Richard Turkington, MD, Principal Investigator — Queens University
Locations (1):
- Belfast City Hospital, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brown M, O'Connor D, Turkington R, Eatock M, Vince R, Hulme C, Bowdery R, Robinson R, Wadsley J, Maraveyas A, Prue G. Feasibility of delivering supervised exercise training following surgical resection and during adjuvant chemotherapy for pancreatic ductal adenocarcinoma (PRECISE): a case series. BMC Sports Sci Med Rehabil. 2023 Sep 21;15(1):116. doi: 10.1186/s13102-023-00722-3. PMID 37735664